CLINICAL TRIAL: NCT00520182
Title: Community Trial to Assess the Effect of Nutritional Intervention Models on Medical Outcomes Among Obese Type 2 Diabetic Patients
Brief Title: Dietary Interventions in Type 2 Obese Diabetic Patients in the Community
Acronym: DIPAC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ben-Gurion University of the Negev (Other)
Collaborators: The S. Daniel Abraham International Center for Health and Nutrition (Other); Clalit Health Services (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RCT3645
Record Dates: First submitted 2007-08-22; First posted 2007-08-23 (Estimated); Last update posted 2007-09-20 (Estimated); Status verified 2007-09

CONDITIONS: Diabetes Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): ADA 2003 diet
  Interventions: Behavioral: ADA 2003
- 2 (Active Comparator): Low Glycemic index (LGI) diet
  Interventions: Behavioral: Low Glycemic index (LGI) diet
- 3 (Active Comparator): MUFA diet
  Interventions: Behavioral: MUFA diet

INTERVENTIONS:
Behavioral: MUFA diet — Patients were advised to consume 23 cal/kg/day. The diet contained sodium (up to 3000mg/day), potassium (more than 3000 mg/day), calcium (around 1300 mg/day) and magnesium (more than 800 mg/day). MUFA diet included only low glycemic index carbohydrates. The diet consisted of 35% carbohydrates and 45% fat (50% of them were mono-unsaturated fatty acids [MUFA]). Participants were advised to eat 4-6 meals per day according to their lifestyle and to participate in 30-45 min of aerobic activity at least 3 days a week.
  Arms: 3
Behavioral: ADA 2003 — Patients were advised to consume 23 cal/kg/day. The diet contained sodium (up to 3000mg/day), potassium (more than 3000 mg/day), calcium (around 1300 mg/day) and magnesium (more than 800 mg/day). The carbohydrates are with mixed glycemic index. The diet contains 50-55% carbohydrates, 30% fat and 15-20% protein. Participants were advised to eat 4-6 meals per day according to their lifestyle and to participate in 30-45 min of aerobic activity at least 3 days a week.
  Arms: 1
Behavioral: Low Glycemic index (LGI) diet — Patients were advised to consume 23 cal/kg/day. The diet contained sodium (up to 3000mg/day), potassium (more than 3000 mg/day), calcium (around 1300 mg/day) and magnesium (more than 800 mg/day). LGI diet included only low glycemic index carbohydrates. The diet consisted of 50-55% carbohydrates, 30% fat and 20%. protein. Participants were advised to eat 4-6 meals per day according to their lifestyle and to participate in 30-45 min of aerobic activity at least 3 days a week.
  Arms: 2

SUMMARY:
Obese patients with type 2 diabetes often fail to loose weight and thus do not succeed in improving their sugar and lipid profiles and remain at high risk for diabetes complications

The study enrolled 259 obese diabetic patients attending HMO clinics in central Israel. Over a 6 month period the participants met with a dietitian every fortnight and attended group lectures every 2 months.

The objective of this intervention was to compare three dietary intervention along with close monitoring of the patients by dietitians, regarding blood lipid and sugar balance as well as weight loss. The three diets are the American Diabetes Association (ADA) diet from 2003; a diet containing low glycemic index carbohydrate otherwise similar to the ADA diet; and a low glycemic index diet with more fat than the other 2 diets with high proportion of mono-unsaturated fatty acids.

Patients were individually randomized to receive one of the three diets. Among the measures obtained every 3 months for the first year and every 6 months thereafter are weight, fasting insulin and glucose, glycosylated hemoglobin, blood and urine chemistry profiles and lipid profile.

ELIGIBILITY:
Inclusion Criteria:

1. Age 30-65years
2. DM2 diagnosed within 1-10 years
3. Body mass index (BMI) 27-34 kg/m²
4. Last HbA1c measurement 7%-10%
5. Last plasma triglyceride (TG) levels 160-400 mg/dl
6. Last serum creatinine less than 1.4 mg/dl
7. No change in diabetes medication for at least three months before entering the study

Exclusion Criteria:

1. Proliferative diabetic retinopathy
2. Current insulin treatment
3. Active oncologic or psychiatric disease
4. Uncontrolled hypothyroidism or hyperthyroidism

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2004-03; Study Completion 2008-02 (Estimated)

PRIMARY OUTCOMES:
Triglyceride level, glycated hemoglobin level, fasting plasma glucose | baseline and every 3 months during year 1, every 6 months therafter

SECONDARY OUTCOMES:
Weight, BMI, waist hip circumference, insulin resistance using HOMA (fasting glucose to fasting insulin ration), HDL-Cholesterol level. | baseline, every 3 months in year 1, every 6 months therafter

CONTACTS AND LOCATIONS:
Overall Officials: Drora Fraser, PhD, Study Chair — Ben-Gurion University of the Negev
Locations (1):
- Clalit HMO, Rehovot, Petach Tikva, Ramle, Central District, Israel

REFERENCES:
- [Result] Shahar DR, Abel R, Elhayany A, Vardi H, Fraser D. Does dairy calcium intake enhance weight loss among overweight diabetic patients? Diabetes Care. 2007 Mar;30(3):485-9. doi: 10.2337/dc06-1564. PMID 17327309
- [Derived] Elhayany A, Lustman A, Abel R, Attal-Singer J, Vinker S. A low carbohydrate Mediterranean diet improves cardiovascular risk factors and diabetes control among overweight patients with type 2 diabetes mellitus: a 1-year prospective randomized intervention study. Diabetes Obes Metab. 2010 Mar;12(3):204-9. doi: 10.1111/j.1463-1326.2009.01151.x. PMID 20151996